CLINICAL TRIAL: NCT03782285
Title: Sacrospinous Ligament Fixation With Conventional Surgical Instruments in Chinese Apical Prolapse Female Patients: a Multi-center Prospective Clinical Trial
Brief Title: Sacrospinous Ligament Fixation With Conventional Surgical Instruments in Chinese Apical Prolapse Female Patients
Acronym: SSLF-CSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: First Hospitals affiliated to the China PLA General Hospital (Other Government); Shanghai First Maternity and Infant Hospital (Other); The Second Hospital of Anhui Medical University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Foshan Women's and Children's Hospital (Other); Suzhou Municipal Hospital (Other); Chongqing Maternal and Child Health Hospital (Other); Hangzhou Maternal and Child Health Hospital (Unknown); Beijing Obstetrics and Gynecology Hospital (Other); Peking Union Medical College (Other); St. Francis Hospital, Chicago, USA (Unknown); University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUnion：SSLF-CSI
Record Dates: First submitted 2018-12-07; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: apical prolapse; sacrospinous Ligament Fixation
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: sacrospinous Ligament Fixation — sacrospinous ligament suspension (SSLF) as a typical native tissue repair procedure is one of the most widely used vaginal procedures for correcting apical prolapse. Ischial spinous fascia fixation (ISFF) will be the replacement procedure if SSLF will not be accomplished by conventional surgical instruments due to unsatisfactory exposure of spinous fascia.
  Other Names: ischial spinous fascia fixation

SUMMARY:
SSLF is typically a suture-based attachment of the vaginal apex to the sacrospinous ligament, either unilaterally or bilaterally. It is usually accomplished with specially designed equipment in English-language scientific literature. However, these instruments either reusable or disposable are relatively expensive and difficult in accessibility, and are not yet widely applied around China. Typical Asian smaller pelvis offers us an optional repair procedure with conventional surgical instruments instead of special instrument.

DETAILED DESCRIPTION:
Apical prolapse is defined as descent of the uterus and cervix, the cervix alone, or the post-hysterectomy vaginal cuff down to the hymen, lower vagina, or past the introitus. Among 684,250 POP procedures that were performed in 15 Organization for Economic Co-operation and Development (OECD) countries in 2012, apical compartment repairs represented 20% of these procedures. Sacrospinous ligament suspension (SSLF) as a typical native tissue repair procedure is one of the most widely used vaginal procedures for correcting apical prolapse. SSLF is typically a suture-based attachment of the vaginal apex to the sacrospinous ligament, either unilaterally or bilaterally usually with specially designed equipment such as Deschamps ligature carrier or Miya hook. However, these instruments are expensive and are not yet widely applied in China. Typical Asian smaller pelvis offers us an optional repair procedure with conventional surgical instruments instead of special instrument. Previous pilot study from Peking Union Medical College Hospital showed promising curative results with conventional surgical instruments in Chinese female patients. The investigation may show us a feasible, economic and effective modified procedure for Asian patients with medium compartment prolapse.

This is a multi-center, prospective clinical trial. Previous studies using conventional surgical instruments for 1-year follow-up showed objective cure rate was 98%, subjective satisfaction was 94%, Considering that the objective cure rate may decrease in multicenter trials, it is assumed that the objective cure rate of multicenter trials can reach 95%. When the sample size is at least 79 patients, 80% of the test efficiency can verify that the objective cure rate is higher than the target value when the bilateral α=0.05. The missing rate was about 10%. The incidence of SSLF failure requiring other operations method due to deep pelvic cavity and unsatisfactory exposure by conventional instruments was about 5%. The final number of cases included in this study should be 100 cases. Ischial spinous fascia fixation (ISFF) will be the replacement procedure if SSLF will not be accomplished by conventional surgical instruments due to unsatisfactory exposure of spinous fascia. The research units will collect perioperative data and complete unified format case report form (CRF) for all selected patients for further analysis. A total of at most 9 months will be required to complete the study after starting up.

ELIGIBILITY:
Inclusion Criteria:

1. Women with apical prolapse with POP-Q III or IV
2. Unilateral (all sutured to right sacrospinous ligament) SSLF is planned，while with vaginal hysterectomy, anterior/posterior vaginal wall repair or mid-urethral suspension could be performed simultaneously.
3. Women who have been eligible for long-term follow-up.
4. Women who agreed to participate in the study and signed informed consent.

Exclusion Criteria:

1. Women who have surgical history for prolapse
2. Women who have contraindication for surgical procedure
3. Women who are unable to comply with the study procedures

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Women with apical prolapse with POP-Q III or IV who are planned to have unilateral SSLF is planned
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-23 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Success rate of SSLF with conventional instruments | up to 36 months after operation
  1. Symptomatic prolapse below grade II occurred at 3 months after operation, and the severest indication point in POP-Q evaluation was taken as the criterion. No vaginal swelling sensation, that is answer "no" for PFDI-20 Questionnaire Question 3, "Do you often see or feel vaginal tumors come out?".
  2. The patient's self-perception symptoms is improved or improved significantly, that is answer 1 or 2 for the PGI-C questionnaire.
  3. There is no need of further treatment for prolapse, such as reoperation or pessary.
  4. Pelvic MRI evaluation on postoperative 3 months follow-up

SECONDARY OUTCOMES:
Postoperative recurrence | from 3 months after operation up to 36 months after operation
  Evaluation on the prolapse of the anterior, middle and posterior pelvic confirms POP-Q II degrees and above.
visual analogue scales | within 3 days after operation
  postoperative pain evaluation esp. hip pain by visual analogue scales (VAS). Visual Analogue Scale (VAS) is a self-report measure consisting simply of a 10 centimeter line with a statement at each end representing one extreme of the dimension being measured (most often intensity of pain)
symptomatic improvement using validated instruments(PFIQ-7) | up to 36 months after operation
  Relief of symptoms using validated instruments, pelvic floor impact questionnaire short form 7(PFIQ-7)。PFIQ-7 scores 0-300, the higher the severer negative influence on patient.
symptomatic improvement using validated instruments(PFDI-20) | up to 36 months after operation
  Relief of symptoms using validated instruments, pelvic floor distress inventory short form 20(PFDI-20), PFDI-20 scores 0-300, the higher the severer negative influence on patient.
symptomatic improvement using validated instruments(PISQ-12) | up to 36 months after operation
  Relief of symptoms using validated instruments, Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire short form(PISQ-12), PISQ-12 scores 0-48, the higher, the severer negative influence on patient.
symptomatic improvement using patient global impression of change (PGI-C) | up to 36 months after operation
  Relief of symptoms using patient global impression of change (PGI-C)， PGI-C scores 1-7, the higher, the the severer negative influence on patient.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Study Chair — Peking Union Medical College Hospital; Yongxian Lu, Principal Investigator — 1st Affiliated hospital of PLA general hospital; Zhiyuan Dai, Principal Investigator — Shanghai First Maternity and Infant Hospital; Wenyan Wang, Principal Investigator — 2nd Affiliated hospital of Anhui Medical college; Zhaoai Li, Principal Investigator — Shan'xi Province Women's and Children's Hospital; Yuling Wang, Principal Investigator — Foshan Women's and Children's Hospital; Shunyu Hou, Principal Investigator — Suzhou City Hospital; Lubin Liu, Principal Investigator — Chongqing Women's and Children's Hospital; Xiangjuan Li, Principal Investigator — Hangzhou Women's and Children's Hospital; Le Ma, Principal Investigator — Beijing Obstetrics and Gynecology Hospital; Tao Xu, Principal Investigator — Statistics Department of Peking Union Medical College; Joseph Schaffer, Principal Investigator — University of Texas Southwestern Medical Center; Marko J Jachtorowycz, Principal Investigator — Saint Francis Hospital
Locations (9):
- China (9):
  - 2nd Affiliated hospital of Anhui Medical college, Hefei, Anhui
  - 1st Affiliated hospital of PLA general hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Women's and Children's Hospital, Chongqing, Chongqing Municipality
  - Foshan Women's and Children's Hospital, Foshan, Guangdong
  - Suzhou City Hospital, Suzhou, Jiangsu
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - Shan'xi Province Women's and Children's Hospital, Taiyuan, Shanxi
  - Hangzhou Women's and Children's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haya N, Baessler K, Christmann-Schmid C, de Tayrac R, Dietz V, Guldberg R, Mascarenhas T, Nussler E, Ballard E, Ankardal M, Boudemaghe T, Wu JM, Maher CF. Prolapse and continence surgery in countries of the Organization for Economic Cooperation and Development in 2012. Am J Obstet Gynecol. 2015 Jun;212(6):755.e1-755.e27. doi: 10.1016/j.ajog.2015.02.017. Epub 2015 Feb 25. PMID 25724403
- [Result] Barber MD, Maher C. Apical prolapse. Int Urogynecol J. 2013 Nov;24(11):1815-33. doi: 10.1007/s00192-013-2172-1. PMID 24142057
- [Result] Ren C, Song XC, Zhu L, Ai FF, Shi HH, Sun ZJ, Chen J, Lang JH. [Prospective cohort study on the outcomes of sacrospinous ligament fixation using conventional instruments in treating stage Ⅲ-Ⅳ pelvic organ prolapse]. Zhonghua Fu Chan Ke Za Zhi. 2017 Jun 25;52(6):369-373. doi: 10.3760/cma.j.issn.0529-567X.2017.06.003. Chinese. PMID 28647958